CLINICAL TRIAL: NCT03826368
Title: Evaluation of Hemp-Derived Botanical Dietary Supplementation to Promote Healthy Brain Function During Recovery From Brain Injury
Brief Title: Hemp-Derived Botanical Dietary Supplementation During Recovery From Brain Injury
Status: Withdrawn | Type: Observational
Why Stopped: Lack of initial funding after approval of study
Sponsor: Real Time Diagnostics Ventures INC (Industry)
Responsible Party: Principal Investigator, Donald Cooper Ph.D., Principal Investigator, Real Time Diagnostics Ventures INC
Other Study IDs: 2018/07/17
Record Dates: First submitted 2019-01-29; First posted 2019-02-01 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Traumatic Brain Injury
Keywords: Cannabinoid; CBD
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Cannabidiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Saliva swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TBI Controls: Adult men and women between 18 and 55. No prior history of traumatic brain injury. Experienced taking hemp-derived botanicals.
  Interventions: Dietary Supplement: Hemp-derived botanical dietary supplement
- TBI HDS: Adult men and women between 18 and 55. History of traumatic brain injury. Experienced taking hemp-derived botanicals.
  Interventions: Dietary Supplement: Hemp-derived botanical dietary supplement

INTERVENTIONS:
Dietary Supplement: Hemp-derived botanical dietary supplement — Subjects currently taking phytocannabinoid Hemp-derived botanical dietary supplements during recovery from brain injury.
  Other Names: Cannabidiol; CBD

SUMMARY:
The objective of the proposed research is to evaluate adult subjects currently taking phytocannabinoid Hemp-derived botanical supplements (HDS) during recovery from traumatic brain injury. This study seeks to answer whether subjects taking HDS formulations experience relief from self-reported symptoms or improved subjective well-being, sleep quality, cognitive benefits, side effects and/or quantifiable changes in brain state neuronal activity or stress biomarkers. We seek to answer whether regular users (once/week to multiple uses/day) of HDS experience signs of dependence, addiction or physiological withdrawal. To accomplish this we will use survey questions, quantitative EEG, cognitive testing and salivary biomarkers to determine the effectiveness of self-initiated HDS administration. In addition, we are interested in whether our objective measures allow us to understand why some people are responders to HDS health benefits while others are not.

ELIGIBILITY:
Inclusion Criteria: Adult male or female volunteers between the ages of 18-55 who have experience a head trauma/ concussion resulting in the diagnosis of mild to moderate TBI (Glasgow Coma scale score between 9-14) with less than 30 minutes of unconsciousness and post-traumatic amnesia lasting less than 24 hours more than 1 month ago will be considered for participation in the study. Volunteers must be able to move about the community of the Denver metro area and speak fluent English. They must be able to leisurely ride a stationary recumbent bicycle without assistance for 10 minutes and sit stationary for 15 minutes without discomfort. They must be familiar with the brand and dosing of HDS and been regular users, defined as once /week up to multiple uses per day for at least 1 month in the past year. They must be able to hear a 25 decibels in at least one ear and respond verbally to questions while remaining still.

Exclusion Criteria:

Medications. Most subjects may continue to take medications for other conditions. However, subjects should be on stable doses of these medications for a specified period prior to beginning the study. A stable dose means that there have been no changes in the drug dosage during the past 2 months.

Subjects may not be current users of illegal drugs (e.g., cocaine, methamphetamine) Subjects may not have an immune-relevant disease (e.g. HIV, MS, Lyme Disease) Females may be pregnant or lactating and taking HDS supplementation. In the consent form we will include a warning that taking cannabis related products during pregnancy or while nursing could pose a danger to the development of the infant.

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults with a history of brain injury and experience taking hemp-derived phytocannabinoid hemp supplements during the recovery period. Controls without brain injury and experience with hemp supplements.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04-13 (Estimated); Primary Completion 2020-04-13 (Estimated); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Symptom inventory | Subjects complete the symptom inventory within 30 minutes of arriving to testing facility after signing the consent forms.
  Sleep and broad symptom inventory
qEEG frequency, brain region coherence assessment baseline measured once immediately after completion of symptom inventory at the testing facility. | Subjects are assessed once immediately after completion of the symptom inventory lasting approximately 10 minutes.
  Frequency power spectral analysis, coherence at baseline in control subjects and treatment group subjects.
qEEG frequency, brain region coherence assessment, pedaling RPM change measured during a 30-40 minute window after baseline testing. | Subjects are assessed once immediately after baseline qEEG test for 30-40 minutes.
  Frequency power spectral analysis, coherence before and after peddling and during memory task where the subject is asked to name or spell the months of the year backwards while pedaling and EEG measurements are taken. Auditory tones are delivered via headsets and the subject is asked to report changes when they detect a change in frequency while attending to a blinking screen.

SECONDARY OUTCOMES:
Subject Accuracy during memory task | Subjects are assessed once immediately after baseline qEEG test for 30-40 minutes.
  Subjects are asked to spell the name of the months or weeks backwards while pedaling a stationary bicycle.

IPD SHARING:
Plan to Share IPD: No